CLINICAL TRIAL: NCT06593132
Title: Prospective Clinical Study of Single Port Endoscopic Breast Conserving Surgery or Open Breast Conserving Surgery for Early Breast Cancer
Brief Title: Single Port Endoscopic Breast Conserving Surgery
Status: Recruiting | Type: Observational
Sponsor: Ren,Yu (Other)
Responsible Party: Sponsor-Investigator, Ren,Yu, chief physician, First Affiliated Hospital Xi'an Jiaotong University
Organization: First Affiliated Hospital Xi'an Jiaotong University (Other)
Other Study IDs: SPEBCS-2023
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Conserving Surgery; Endoscopic Surgery
Keywords: breast conserving surgery; single port endoscopic; early breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- single port endoscopic breast conserving surgery: Endoscopic breast conserving surgery, which uses breast endoscope for breast conserving surgery, can not only preserve the breast completely, but also meet the appearance needs of patients with breast preservation, and has more advantages than traditional surgery.
  Interventions: Procedure: endoscopic breast conserving surgery
- open breast conserving surgery: On the surface of the breast tumor centered, is apart from the 2 cm do arc, radial incision tumor, tags in the cut edge around the joints and removing tissue inspection, to ensure the cut edge negative.
  Interventions: Procedure: endoscopic breast conserving surgery

INTERVENTIONS:
Procedure: endoscopic breast conserving surgery — Breast endoscopy technology completes complex surgical operations through small incisions, achieving aesthetically pleasing results while ensuring tumor safety.

SUMMARY:
The center plans to carry out a prospective clinical study of single hole total endoscopic breast conserving surgery for early breast cancer compared with open breast conserving surgery, to provide high-level evidence-based medical evidence for the development of endoscopic breast conserving surgery for early breast cancer.

DETAILED DESCRIPTION:
Data show that breast cancer has surpassed lung cancer asthemost prevalent malignant tumor in the world, and traditional open surgery is highly invasive and has poor cosmetic results. This study investigates the results of endoscopic breast- conserving surgery(E-BCS) versus conventional breast-conserving surgery(C-BCS) in the treatment of patients with early-stage breast cancer and to compare the advantages and disadvantages of the two surgical procedures, so as to provide the best evidence for the rational choice of the procedure by both doctors and patients.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer confirmed by pathology；
2. Tumor <5 cm, TNM stage 0-II；
3. Single Port Endoscopic or traditional open surgery; (4)20 to 70 years old female patients.

Exclusion Criteria:

1. Bilateral breast cancer;
2. Reconstruction after breast conserving surgery ;
3. Basic information is not complete；
4. Breast conserving surgery was converted to modified radical resection or subcutaneous adenoidectomy.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants are women
Study Population: Female patients aged 20-70 years who are eligible for breast-conserving surgery and are willing to undergo breast-conserving surgery.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Six months after operation SURVIVAL EFFECTS | From enrollment to the end of 6 months after surgery
  To compare the overall survival (OS) within 6 months after single-port endoscopic breast-conserving surgery and open breast-conserving surgery.

SECONDARY OUTCOMES:
Intraoperative blood loss | From the beginning to the end of the operation
  To compare the total blood loss between single-port endoscopic breast-conserving surgery and open breast-conserving surgery.
Postoperative drainage volume in the first three days after breast conserving surgery | 3 days after surgery
  The total drainage volume in the first three days after breast conserving surgery was compared between single-port endoscopic breast conserving surgery and open breast conserving surgery.
Length of surgical incision | 1 week after surgery
  The total incision length was compared between single-port endoscopic breast-conserving surgery and open breast-conserving surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No